CLINICAL TRIAL: NCT05188703
Title: Undiagnosed Diabetic Retinopathy: Using Participatory Science to Design an Intervention for Patients at High-Risk for Blindness
Brief Title: Patient Navigator Intervention for Diabetic Retinopathy
Acronym: SEEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000031731; 1K23EY030530-01 (NIH)
Record Dates: First submitted 2021-12-22; First posted 2022-01-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Retinopathy; Diabetic Blindness
Keywords: diabetic retinopathy; diabetic blindness; patient navigator
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: This is a single arm study. All participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Intervention consists of standard of care eye exam and enrollment in a patient navigation program.
  Interventions: Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Patient Navigation — Participants will be assigned to a patient navigator and will have quarterly appointments. Patient navigators will assist with access and coordination of medical care.

SUMMARY:
This is a pilot study of a patient navigator intervention for people living with diabetes and at high risk of diabetic blindness. The investigators are assessing the feasibility and acceptability of the intervention in preparation for a clinical trial.

DETAILED DESCRIPTION:
Evidence-based treatment for Diabetic retinopathy (DR) established 30 years ago decreases the likelihood of blindness by 50%. Outcomes are even better now with emerging therapies and technology. Diabetes remains the leading cause of new cases of legal blindness. This study is significant because it investigates the gap between published guidelines and the population that continues to go blind despite well-established recommendations for screening. Our current model of screening for DR screens much of the population appropriately. There is an opportunity to improve DR screening by timely identification of persons at risk for preventable blindness. DR disproportionately impacts Non-Hispanic Blacks, Latinos, Native Americans, and lower socioeconomic communities. Racial and ethnic minorities are less likely to be screened for DR, have a higher prevalence of disease, and more severe disease. There is not a clear path toward decreasing these disparities beyond these data. This study addresses barriers to the implementation of evidenced-based treatment protocols by identifying modifiable patient and population-level challenges and building an intervention informed by community members and national data. It is a direct response to the "population health imperative" described by the National Academies of Science, Engineering, and Medicine. Our study answers the National Eye Institute's Strategic Plan request to evaluate disparities by identifying barriers that prevent optimal treatment. It is aligned with the NEI's mission to support research and training with respect to the preservation of sight. The National Institute on Minority Health and Health Disparities Research Framework provides the conceptual foundation for our work. Our proposal identifies facets of the biologic, built, and sociocultural environments of the national population with undiagnosed DR. The national analysis informs a local individual-level intervention that addresses determinants associated with DR screening. The scientific premise of this study is the forty percent of persons with diabetes not screened despite established sight-saving treatment, the known disparities in screening for DR, and the increased prevalence of sight-threatening DR in Black, Latino, Native, and lower income Americans.

Primary Objective The primary objective of this study is to design and pilot a patient navigator program to increase screening for DR in a high-risk population.

Secondary Objective To determine the feasibility and accessibility of a patient navigation program for persons at high-risk for DR.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Diagnosis of diabetes and record of diagnosis in YNHHS EPIC
* English-speaking
* No documented eye examination within 1 year of study enrollment
* High risk for diabetic retinopathy based on risk calculator evaluation

Exclusion Criteria:

* Documented eye exam in the past year
* Not high risk for diabetic retinopathy
* Diabetes diagnosis not recorded in EPIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Number of participant who had baseline eye exam | 18 months
  The number of participants who had their baseline eye exam will be determined using the electronic health record
Number of participants who completed a follow-up eye exam 12+ months after baseline eye exam | up to 18 month
  The number of participants who completed a follow-up eye exam 12+ months after baseline eye exam will be determined using the electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nwanyanwu, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make IPD available to other researchers.

REFERENCES:
- [Background] Nwanyanwu KMJH, Nunez-Smith M, Gardner TW, Desai MM. Awareness of Diabetic Retinopathy: Insight From the National Health and Nutrition Examination Survey. Am J Prev Med. 2021 Dec;61(6):900-909. doi: 10.1016/j.amepre.2021.05.018. Epub 2021 Aug 21. PMID 34426057